CLINICAL TRIAL: NCT02550561
Title: Pilot Study of Percutaneous Posterior Tibial Nerve Stimulation for the Treatment of Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: Pilot Study of Percutaneous Posterior Tibial Nerve Stimulation for the Treatment of IC/PBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Felicia Lane, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-2010
Record Dates: First submitted 2015-09-03; First posted 2015-09-15 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: Posterior tibial nerve stimulation; PTNS; IC
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Posterior Tibial Nerve Stimulation (Experimental): PTNS (under the brand name Urgent PC) is an FDA-approved device for the treatment of urinary urgency, urinary frequency and urge incontinence. It is often described as a peripheral form of neuromodulation (as opposed to SNM which is central neuromodulation at the level of the nerve root). PTNS involves 12 weeks of weekly 30 minute office-based treatment sessions with a small electrode placed slightly above the ankle in order to stimulate the S2-4 nerve roots. If benefits are obtained, 12 weeks of treatment is followed by spaced maintenance sessions at timing of provider and patient discretion.
  Interventions: Device: Posterior Tibial Nerve Stimulation

INTERVENTIONS:
Device: Posterior Tibial Nerve Stimulation — PTNS (under the brand name Urgent PC) is an FDA-approved device for the treatment of urinary urgency, urinary frequency and urge incontinence. It is often described as a peripheral form of neuromodulation (as opposed to SNM which is central neuromodulation at the level of the nerve root). PTNS involves 12 weeks of weekly 30 minute office-based treatment sessions with a small electrode placed slightly above the ankle in order to stimulate the S2-4 nerve roots.

SUMMARY:
In 2014, the American Urological Association updated it management algorithm for Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS). As the algorithm progresses, interventions become increasingly invasive and morbid. 4th line treatment is sacral neuromodulation (SNM), involving a two stage surgical procedure and permanent device implantation. While the mechanism for decrease in IC/PBS symptoms is unknown, SNM is thought act through central and peripheral mechanisms related to afferent signaling, causing modification of pain and lower urinary tract sensation.¹

Percutaneous posterior tibial nerve stimulation (PTNS) is a method of peripheral neuromodulation targeting the same nerve roots as SNM, but with significantly fewer risks. The purpose of our research is to determine if PTNS is effective in the treatment of IC/PBS. The results of this study will suggest future directions and provide critical information to design studies to determine to what extent and in what situations PTNS may be effective.

The investigators will enroll subjects with IC/PBS and urinary frequency/urgency to treatment with 12 weekly treatments of PTNS. The investigators will assess symptoms and lower urinary tract function before, during and after the treatments. At the completion of treatments, subjects will be asked to enroll in post-study follow up monitoring to understand the duration of symptom effect.

DETAILED DESCRIPTION:
The overall objective of this prospective, pilot study is to determine if percutaneous tibial nerve stimulation (PTNS) is an effective treatment for interstitial cystitis/painful bladder syndrome (IC/PBS). Our specific aim is to evaluate how PTNS performs with regards to the reduction of symptoms in subjects with this disorder. The primary outcome variable will be the percentage of subjects to report that they are moderately improved or markedly improved in overall symptoms compared to baseline on a 7-point global response assessment (GRA) scale. The GRA scale involves asking the question, "As compared to when you started the current study, how would you rate your overall symptoms now?". There are 7 possible responses: markedly worse, moderately worse, slightly worse, the same, slightly improved, moderately improved and markedly improved. This scale is the current standard for outcome in studies that are evaluating treatments and interventions for IC/PBS.

There will be a number of secondary outcome variables including: changes in a 24 hour voiding diary during the course of the interventions, ratings for bladder pain, urinary urgency and urinary frequency on standardized scales, the score on O'Leary-Sant IC Symptom and Problem Index, scores of validated questionnaires for pelvic floor and general health. The investigators will also collect and report any adverse events.

Subjects will be recruited during a routine visit to the University of California, Irvine (UCI) urogynecology division that the patient has scheduled to initiate or continue routine care for their complaints. If the provider feels that the patient may be appropriate for the study and meets the inclusion/exclusion criteria, she will offer to have a study investigator speak with patient at that time or at a later time at the patient's convenience. Once consents are signed, the subject will be provided with the following materials to complete before their first treatment visit:

1. demographic and medical history survey
2. 24 hour voiding diary
3. visual analog scale (VAS) for bladder pain
4. Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF Questionnaire)
5. O'Leary-Sant IC Symptom and Problem Index
6. urine pregnancy test (for premenopausal subjects)

The PTNS treatment visits will be administered in the standard fashion. This involves the placement of a thin needle (similar to an acupuncture needle) inserted near the posterior ankle. The needle is then connected to an electrode stimulator and the stimulation is adjusted until appropriate response (toe flex or fan) is obtained without patient discomfort. When at the appropriate level, the electrode is stimulated for 30 minutes per treatment session.

Study visits will be conducted in the UCI Ob/Gyn clinic with a nurse trained to administer PTNS. These treatments will occur weekly for 12 weeks. (See Section 2.4 for table outlining treatment visits.) At all visits, the nurse will inquire regarding any adverse reactions to treatment and the subject complete a VAS. After completion of the twelfth treatment visit, the subject will be requested to complete the following:

1. 7-point global response assessment (GRA) scale and interval medical history questionnaire
2. 24 hour voiding diary
3. visual analog scale (VAS) for bladder pain
4. Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF Questionnaire)
5. O'Leary-Sant IC Symptom and Problem Index

These forms will be returned within two weeks and the subject will return to the clinic for a follow up visit with her provider. At this time, depending on their current symptoms and response to the treatment on the GRA scale, the subjects will be offered to continue with PTNS treatments at a maintenance interval or to pursue alternative care outside of the study protocol if no benefit was obtained. If subjects are planning to continue maintenance treatments, they will be asked if they wish to continue with an additional follow up 12-16 weeks after the final treatment visit. The information collected at that time will be as follows:

1. 7-point global response assessment (GRA) scale and interval medical history questionnaire
2. 24 hour voiding diary
3. visual analog scale (VAS) for bladder pain
4. Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF Questionnaire)
5. O'Leary-Sant IC Symptom and Problem Index
6. Post-study follow-up survey

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of IC/PBS
* complaint of urinary urgency (sudden, compelling desire to pass urine which is difficult to defer) or urinary frequency (voiding >8 times per 24 hour period)
* female
* have undergone at least 1 course of a standard therapy for IC/PBS
* 18 years of age or older

Exclusion Criteria:

* not having undergone at least 1 course of a standard therapy for IC/PBS
* having a pacemaker or implantable defibrillator
* being prone to excessive bleeding
* having nerve damage that could impact the posterior tibial nerve
* pregnant or planning pregnancy during treatment course
* non-English speaking
* current malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California-Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posterior Tibial Nerve Stimulation
Started | 16
Completed | 10
Not Completed | 6
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Posterior Tibial Nerve Stimulation
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 16
VAS score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (VAS) ranges from 0 to 10 with higher values representing a worse outcome.
  units on a scale | 4.2 (2.3)
Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) questionnaire score [Mean (Standard Deviation); unit: units on a scale] — The Pelvic Pain and Urgency/Frequency Patient Symptom Scale contains the sum of symptom and bother scores. There is a total of 8 questions but, due to sub-questions, there are 11 answers about severity of condition coded in a range from 0 to 4 subscale for two questions and 0 to 3 for nine questions. Scores with higher values represent a worse outcome. The total score sum is reported and ranges from 0 to 35.
  units on a scale | 17.5 (5.9)
O'Leary-Sant IC Symptom Index (ICSI) score [Mean (Standard Deviation); unit: units on a scale] — O'Leary-Sant Interstitial Cystitis Symptom Index score is a sum of responses ranging from 0 to 5 for four questions, totaling from 0 to 20. Higher values represent worse outcome.
  units on a scale | 11.2 (4.2)
O'Leary-Sant IC Problem Index (ICPI) score [Mean (Standard Deviation); unit: units on a scale] — O'Leary-Sant Interstitial Cystitis Problem Index score is a sum of responses ranging from 0 to 4 for four questions, totaling from 0 to 16. Higher values represent worse outcome.
  units on a scale | 10.2 (3.7)
24 hour voiding frequency [Mean (Standard Deviation); unit: voids/24 hours] — The amount of voids in a 24 hour period.
  voids/24 hours | 12.2 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure: Percentage of Subjects Improved Global Response Assessment Scale
Description: The primary outcome variable will be the percentage of subjects to report that they are moderately improved or markedly improved in overall symptoms compared to baseline on a 7-point global response assessment (GRA) scale. The GRA scale involves asking the question, "As compared to when you started the current study, how would you rate your overall symptoms now?". There are 7 possible responses: markedly worse, moderately worse, slightly worse, the same, slightly improved, moderately improved and markedly improved. This scale is the current standard for outcome in studies that are evaluating treatments and interventions for IC/PBS. Responders are those that marked either moderately or markedly improved.
Time Frame: Visit 6 at 6 weeks and Visit 12 at 12 weeks
Population: A total of 21 patients met eligibility for enrollment. 16 subjects enrolled and began treatment with PTNS. Ten subjects completed 12 sessions while six patients were lost to follow up. Of those who were lost to follow up, only one case withdrew due to bladder worsening pain after four sessions
Measure: Count of Participants; unit: Participants
Arm/Group | Posterior Tibial Nerve Stimulation
Number analyzed (Participants) | 10
Participants
  Responders by Visit 6 | 4
  Responders by Visit 12 | 3
Statistical Analysis 1: Comparison: Posterior Tibial Nerve Stimulation; Test type: Superiority; p = 0.317, McNemar — Subjects that reported either moderately or markedly improved on the GRA scale at 6 weeks compared to 12 weeks

2. Secondary Outcome: Composite Secondary Self-Reported Outcome Measures - Questionnaires
Description: Scores with higher values represent a worse outcome for all measures. (1) Visual Analog Scale (VAS) rating of the severity of pain ranges from 0-10; (2) Pelvis Pain and Urgency/Frequency Patient Symptom (PUF) Scale is the sum of symptom and bother scores. There is a total of 8 questions but, due to sub-questions, there are 11 answers about severity of condition coded in a range from 0 to 4 subscale for two questions and 0 to 3 for nine questions. The total score sum is reported and ranges from 0 to 35; (3) O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) score is a sum of responses ranging from 0 to 5 for four questions, totaling from 0 to 20;. (4) O'Leary-Sant Interstitial Cystitis Problem Index (ICPI) score is a sum of responses ranging from 0 to 4 for four questions from 0 to 16.
Time Frame: At baseline then validated at follow-up (12-14 weeks)
Population: Questionnaire means and standard deviations was analyzed and reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Posterior Tibial Nerve Stimulation - Week 6 Score: Scores and standard deviations for questionnaires and 24 hour voiding frequency by participants by week 6.
- Posterior Tibial Nerve Stimulation Week 12: Scores and standard deviations for questionnaires and 24 hour voiding frequency by participants by week 12.
Arm/Group | Posterior Tibial Nerve Stimulation - Week 6 Score | Posterior Tibial Nerve Stimulation Week 12
Number analyzed (Participants) | 10 | 10
score on a scale
  Visual Analog Scale (VAS) | 3.4 (2.2) | 3.2 (2.0)
  Pelvis Pain and Urgency/Frequency Patient Symptom Scale (PUF) | 15.5 (4.7) | 16.1 (3.7)
  O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) | 8.3 (3.8) | 7.8 (3.6)
  O'Leary-Sant Interstitial Cystitis Problem Index (ICPI) | 8.3 (4.3) | 8.6 (3.6)
Statistical Analysis 1: Comparison: Posterior Tibial Nerve Stimulation Week 12; The mean change in Visual Analog Scale (VAS) score for bladder pain; Test type: Other; p = 0.47, paired t-tests
Statistical Analysis 2: Comparison: Posterior Tibial Nerve Stimulation Week 12; The mean change in Pelvis Pain and Urgency/Frequency Patient Symptom (PUF) score; Test type: Other; p = 0.17, paired t-test
Statistical Analysis 3: Comparison: Posterior Tibial Nerve Stimulation Week 12; The mean change for O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI); Test type: Other; p = .08, paired t-test
Statistical Analysis 4: Comparison: Posterior Tibial Nerve Stimulation Week 12; The mean change O'Leary-Sant Interstitial Cystitis Problem Index (ICPI); Test type: Other; p = 0.51, paired t-test
Statistical Analysis 5: Comparison: Posterior Tibial Nerve Stimulation Week 12; The mean change in 24-h urinary frequency; Test type: Other; p = 0.22, paired t-test

3. Secondary Outcome: Secondary Self-Reported Outcome Measures - 24 Hour Voiding Frequency
Description: Scores with higher values represent a worse outcome for all measures. 24-Hour Voiding Diary includes frequency, fluid intake and void amount (ounces), leaks or accidents (yes or no), strong urge to urinate (yes or no), activity when you leaked or had an urge (description)
Time Frame: At baseline then validated at follow-up (12-14 weeks)
Population: Means and standard deviations along with 24-h voiding frequency was analyzed and reported.
Measure: Mean (Standard Deviation); unit: number of voids
Groups:
- Posterior Tibial Nerve Stimulation - Week 6 Score: Scores and standard deviations for 24 hour voiding frequency by participants by week 6.
- Posterior Tibial Nerve Stimulation Week 12: Scores and standard deviations for 24 hour voiding frequency by participants by week 12.
Arm/Group | Posterior Tibial Nerve Stimulation - Week 6 Score | Posterior Tibial Nerve Stimulation Week 12
Number analyzed (Participants) | 10 | 10
number of voids | 10.3 (5.0) | 11.6 (5.4)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected over the period of 12 weeks of PTNS treatment.
Description: Definitions did not differ.
Arm/Group | Posterior Tibial Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT02550561/Prot_SAP_000.pdf